CLINICAL TRIAL: NCT01098838
Title: A Phase I, Multi-center, Open-label, Dose-escalation Study of Oral LCL161 in Adult Patients With Advanced Solid Tumors
Brief Title: Safety and Efficacy of LCL161 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCL161A2101
Record Dates: First submitted 2010-04-01; First posted 2010-04-05 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-08

CONDITIONS: Advanced Solid Tumors
Keywords: Cancer; adults; solid tumor; apoptosis; programmed cell death; LCL161
MeSH Terms: conditions — Neoplasms | interventions — LCL161

ARMS (3):
- Weekly dosing of LCL161 (Experimental): by mouth (oral)
  Interventions: Drug: LCL161
- Comparison of LCL161 (Experimental): tablet versus liquid
  Interventions: Drug: LCL161
- Twice daily dosing of LCL161 (Experimental): by mouth for 4 days followed by a 3-day rest period every week
  Interventions: Drug: LCL161

INTERVENTIONS:
Drug: LCL161

SUMMARY:
The study will evaluate the safety of increasing doses of oral LCL161 in patients with solid tumors. It is primarily designed to evaluate the side effects and find the maximum tolerated dose of LCL161.

ELIGIBILITY:
Inclusion Criteria:

* Solid tumor
* ECOG performance status 0-2
* Life expectancy greater than or equal to 12 weeks
* Must meet certain blood laboratory values
* Must meet criteria for time since the last dose of prior therapy
* Must provide written informed consent to participate in this study

Exclusion Criteria:

* Active and/or symptomatic brain tumors or brain metastases.
* Patients with unresolved nausea, vomiting, or diarrhea
* Any ongoing severe and/or uncontrolled medical condition that could compromise participation in the study including heart, lung or inflammatory disease
* Any disease that may significantly alter the absorption of the study drug (for example, ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or removal of small bowel)
* Patients who are currently receiving treatment with steroids at a certain dose or other immunosuppressive treatment that cannot be stopped prior to starting study drug
* Patients who are currently receiving treatment with certain medications
* Patients who have received radiation therapy or have undergone major surgery within the last 4 weeks
* Women of child-bearing potential who are pregnant or breast feeding.
* Known diagnosis of human immunodeficiency virus (HIV) infection or chronic active hepatitis B or C
* Patients unwilling or unable to follow the protocol

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2008-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of dose-limiting toxicities | Cycle 1

SECONDARY OUTCOMES:
Frequency and type of adverse events | throughout the study
Comparison of amount of LCL161 that gets into blood stream from tablet formulation versus liquid formulation (bioavailability) | 3 months
Blood assessments to determine how much LCL161 gets into the blood stream (pharmacokinetic parameters) | 4 weeks
Pharmacodynamic measurements to determine how LCL161 interacts with proteins related to cancer such as cIAP, cytokines, and cell death markers; hair, skin and tumor samples will be evaluated for target inhibition | Intermittent throughout treatment period
Solid tumor response criteria will be used to identify any anti-tumor activity | After a minimum of 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- United States (3):
  - UNC/ Lineberger Comprehensive Cancer Center Dept. of LinbergerCancerCtr(2), Chapel Hill, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute DeptofSarahCannonRes.Inst. (2), Nashville, Tennessee

REFERENCES:
- [Derived] Infante JR, Dees EC, Olszanski AJ, Dhuria SV, Sen S, Cameron S, Cohen RB. Phase I dose-escalation study of LCL161, an oral inhibitor of apoptosis proteins inhibitor, in patients with advanced solid tumors. J Clin Oncol. 2014 Oct 1;32(28):3103-10. doi: 10.1200/JCO.2013.52.3993. Epub 2014 Aug 11. PMID 25113756
- See also: Related Info — http://www.NovartisClinicalTrials.com